CLINICAL TRIAL: NCT00443677
Title: Treatment of Advanced Hodgkin's Disease (Stages IIB-III-IV)
Acronym: HD2000
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: sponsor, Gruppo Italiano Studio Linfomi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD2000
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Advanced Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- abvd (Active Comparator)
  Interventions: Drug: COPPEBVCAD vs BEACOPP vs ABVD
- beacopp (Experimental)
  Interventions: Drug: COPPEBVCAD vs BEACOPP vs ABVD
- coppebvcad (Experimental)
  Interventions: Drug: COPPEBVCAD vs BEACOPP vs ABVD

INTERVENTIONS:
Drug: COPPEBVCAD vs BEACOPP vs ABVD

SUMMARY:
The purpose of this study is to compare the toxicities of the COPPEBVCAD vs BEACOPP vs ABVD regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of Hodgkin disease
* Clinical stage IIB, III, IV
* No prior treatment for Hodgkin disease or other malignancy
* Age 18-65 year
* Good cardiac, pulmunar, renal and hepatic function
* Performance status 0-3 (Karnofsky 100- 40)
* Written Informed Consent

Exclusion Criteria:

* HIV positivity
* Large cell, anaplastic, CD30+ lymphoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2000-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To compare the toxicity of the COPPEBVCAD vs BEACOPP vs ABVD regimens

SECONDARY OUTCOMES:
To compare the results in terms of response, failure free survival and relapse free survival of the three regimens

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gobbi, MD, Principal Investigator — GISL; Emilio Iannitto, MD, Principal Investigator — GISL; Giuseppe Polimeno, MD, Principal Investigator — GISL
Locations (1):
- Centro Oncologico Modenese, Modena, Italy